CLINICAL TRIAL: NCT04345679
Title: Anti COVID-19 Convalescent Plasma Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orthosera Kft. (Other)
Collaborators: Semmelweis University (Other); University of Pecs (Other); Hungarian National Blood Service (Unknown); Humán Bioplazma Kft - Kedrion (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AntiCOVID19ORT
Record Dates: First submitted 2020-04-11; First posted 2020-04-14 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: COVID 19
Keywords: COVID-19; convalescent plasma; serum therapy
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hospitalized patients with SARS CoV-2 infection (Experimental)
  Interventions: Biological: anti-SARS-CoV-2 convalescent plasma

INTERVENTIONS:
Biological: anti-SARS-CoV-2 convalescent plasma — Infusion of one unit of anti-SARS-CoV-2 convalescent plasma ~200 mL over 4 hours

SUMMARY:
Why is the research needed? The pandemic known as COVID-19 is now spreading across the world with currently (April 10, 2020) more than 1 115 530 active cases and 96 791 deaths. In most affected countries the current goal is to 'flatten the curve' of the epidemic since there is no health care system that is able to treat an extremely high volume of patients all at once. There is a need for immediately applicable treatments for the patients at highest risk, which gains time until targeted therapies become available. A key feature in the pathomechanism of the disease is that the virus elicits an immunological over-reaction in the human body termed 'cytokine storm'. In susceptible patients this hyper-inflammation itself is a significant burden and may even inhibit the body to generate antibodies against the virus in adequate quantities. Therefore, identifying the subset of patients with excess cytokine response and supplementing them with convalescent plasma from recovered donors may be a life-saving treatment option.

What is our study about? In light of recent promising data on plasma therapy in the treatment of COVID-19 and other viral epidemics, there is a need for better understanding the cytokine response to the virus in order to better characterize the target population for convalescent plasma therapy.

Our hypothesis is that convalescent plasma transfusion from healthy donors who recovered from SARS CoV-2 is able to reduce the cytokine storm in addition to replenish the patient's own antibodies in the acutely infected phase of the disease.

A plasmapheresis donation of 400ml will be performed in subjects who recovered from COVID-19 and who are otherwise eligible for plasma donation. The sample will be tested for anti-SARS CoV-2 neutralizing antibody titers and those that reach the level of 1:320 will be processed for transfusion at the Hungarian National Transfusion Service.

Recipients will be COVID-19 patients requiring hospitalization regardless of the severity of the disease or other co-morbidities. A blood-type matched transfusion of 200 ml convalescent plasma will be infused in a single sitting through an iv. infusion of 4 hours.

Recipients will be followed up at days 1, 3,7,12, 17, 28 for clinical symptoms, antibody levels and cytokine response.

ELIGIBILITY:
Inclusion criteria for blood donors :

* age : >18 and <60 years
* body weight : >50 kg
* confirmed previous SARS CoV-2 infection
* 2 negative SARS CoV-2 test result
* written informed consent
* neutralizing antibody titer min. 1 : 120

Exclusion criteria for blood donors :

* age : <18 or >60 years
* female subjects who are pregnant
* HIV1,2 hepatitis B,C or syphilis infection

to minimize the transfusional side effects our aim is to include mostly male donors.

Inclusion criteria for patients/recipients :

* age : >18 years
* admitted to hospital due to SARS CoV-2 infection
* written informed consent

Exclusion criteria for patients/recipients :

* age : <18 years
* female subjects who are pregnant or breastfeeding
* patients with prior allergic reaction to transfusion
* patients who received in the past 30 days immunoglobulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Changing of viral load of SARS-CoV2 | Day 1,3, 7, 12
  Copies of COVID-19 per ml

SECONDARY OUTCOMES:
Changes in immunglobulin G COVID-19 antibody titer | 12 days
  Immunoglobulin G COVID-19 antibodies Immunglobulin G antibody titer
Changes at the cytokine pattern | 12 days
Intensive Care Unit Admission | Day 7,12,28
  Proportion of patients with Intensive Care Unit Admission requirement
Length of hospital stay | Day 7, 12, 28
  Days of Hospitalization
Duration of mechanical ventilation | Day 7, 12, 28
  Days with mechanical ventilation
Clinical Status | Day 7, 12, 28
  Clinical status assessed according to the World Health Organization guideline
Mortality | Day 7, 12, 28
  Proportion of death patients at days

CONTACTS AND LOCATIONS:
Overall Officials: Veronika Müller, MD, PhD, Principal Investigator — Semmelweis University
Locations (1):
- Semmelweis University's Department of Pulmonology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Belyakov IM, Hel Z, Kelsall B, Kuznetsov VA, Ahlers JD, Nacsa J, Watkins DI, Allen TM, Sette A, Altman J, Woodward R, Markham PD, Clements JD, Franchini G, Strober W, Berzofsky JA. Mucosal AIDS vaccine reduces disease and viral load in gut reservoir and blood after mucosal infection of macaques. Nat Med. 2001 Dec;7(12):1320-6. doi: 10.1038/nm1201-1320. PMID 11726972
- [Background] Arabi Y, Balkhy H, Hajeer AH, Bouchama A, Hayden FG, Al-Omari A, Al-Hameed FM, Taha Y, Shindo N, Whitehead J, Merson L, AlJohani S, Al-Khairy K, Carson G, Luke TC, Hensley L, Al-Dawood A, Al-Qahtani S, Modjarrad K, Sadat M, Rohde G, Leport C, Fowler R. Feasibility, safety, clinical, and laboratory effects of convalescent plasma therapy for patients with Middle East respiratory syndrome coronavirus infection: a study protocol. Springerplus. 2015 Nov 19;4:709. doi: 10.1186/s40064-015-1490-9. eCollection 2015. PMID 26618098
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Kardos D, Marschall B, Simon M, Hornyak I, Hinsenkamp A, Kuten O, Gyevnar Z, Erdelyi G, Bardos T, Paukovits TM, Magos K, Beres G, Szenthe K, Banati F, Szathmary S, Nehrer S, Lacza Z. Investigation of Cytokine Changes in Osteoarthritic Knee Joint Tissues in Response to Hyperacute Serum Treatment. Cells. 2019 Aug 3;8(8):824. doi: 10.3390/cells8080824. PMID 31382623
- [Background] Nacsa J, Edghill-Smith Y, Tsai WP, Venzon D, Tryniszewska E, Hryniewicz A, Moniuszko M, Kinter A, Smith KA, Franchini G. Contrasting effects of low-dose IL-2 on vaccine-boosted simian immunodeficiency virus (SIV)-specific CD4+ and CD8+ T cells in macaques chronically infected with SIVmac251. J Immunol. 2005 Feb 15;174(4):1913-21. doi: 10.4049/jimmunol.174.4.1913. PMID 15699118
- See also: 12. Ethics of using convalescent whole blood and convalescent plasma during the Ebola epidemic. Interim guidance for ethics review committees, researchers, national health authorities and blood transfusion services. 2015 WHO/HIS/KER/GHE/15.1 — http://apps.who.int/iris/bitstream/handle/10665/161912/WHO_HIS_KER_GHE_15.1_eng.pdf;jsessionid=F7C13F58F53ADE7D203B12781D96CF02?sequence=1